CLINICAL TRIAL: NCT00202254
Title: 'Functioning and Disability' and 'Quality of Life' in an Australian Community Cohort With Multiple Sclerosis.
Brief Title: Multiple Sclerosis Rehabilitation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Melbourne Health (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HREC 2004.101; MelbUni HREC 040334
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Multiple Sclerosis
Keywords: Mulitple Sclerosis; MS
MeSH Terms: conditions — Multiple Sclerosis | interventions — Physical Therapy Modalities; Occupational Therapy

INTERVENTIONS:
Behavioral: Physiotherapy
Behavioral: Occupational therapy
Behavioral: Speech pathology

SUMMARY:
The effects of routine rehabilitation in MS patients versus no rehabilitation.

DETAILED DESCRIPTION:
Routine rehabilitation inervention in patients with MS. This comprises of medical and nursing input, physiotherapy, occupational therapy, speech pathology, neuropsychology, compared with a "control" group on the waiting list for rehabilitation intervention. Duration of intervention is 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of MS (Paty)- Community dwelling participants with known neurological and psychological deficits per EDSS groups.- Age 19-64 years.- Male and female participants.- Residing within 60kms of metropolitan Melbourne.- Have mobility problem.- Adequate cognition (KFS=2).

Exclusion Criteria:

* Patients residing in nursing home and other residential care.- Those with severe cognitive problems KFS>2.-

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100
Dates: Start 2004-12; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Improvement in fatigue levels and psychological well being (depression, stress and anxiety) in MS patients. Outcome will be measured at 13 months since recruitment.

SECONDARY OUTCOMES:
- Improvement in function and activities of daily living ie. disability- Quality of life.- Carer Burder in multiple sclerosis.- Utilisation of health services.- 13 months follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Fary Khan, Principal Investigator — Melbourne Extended Care Rehabilitation Service